CLINICAL TRIAL: NCT01833832
Title: Phase II Trial of Surgical Resection and Heated Intraperitoneal Peritoneal Chemotherapy (HIPEC) for Adrenocortical Carcinoma
Brief Title: Surgery and Heated Chemotherapy for Adrenocortical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeremy Davis, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130114; 13-C-0114
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Adrenocortical Carcinoma; Peritoneal Carcinomatosis
Keywords: Synergy for Cisplatin and Hyperthermia; Rare Tumor; Poor Prognosis
MeSH Terms: conditions — Adrenocortical Carcinoma; Peritoneal Neoplasms; Hyperthermia | interventions — Cisplatin; Cytoreduction Surgical Procedures; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cytoreductive surgery followed by HIPEC (Experimental): Cytoreductive surgery followed by hyperthermic intraperitoneal chemotherapy (HIPEC) with cisplatin
  Interventions: Drug: Cisplatin; Procedure: Cytoreductive surgery; Drug: sodium thiosulfate

INTERVENTIONS:
Drug: Cisplatin — Patients who are successfully debulked will then undergo hyperthermic intraperitoneal chemotherapy (HIPEC) with cisplatin.
  Other Names: Platinol
Procedure: Cytoreductive surgery — Patients will undergo cytoreductive surgery to achieve a Completeness of Cytoreduction Score (CC) of 0 or 1.
Drug: sodium thiosulfate — sodium thiosulfate will be given to limit the toxicity of cisplatin

SUMMARY:
Background:

- Adrenocortical carcinoma (ACC) is a rare tumor of the adrenal gland. Few people who develop this disease live more than 5 years after being diagnosed. Those whose tumors have spread inside their abdomen may have an especially poor outcome. In these cases, traditional chemotherapy is not very effective. One possible new treatment is aggressive surgery with heated chemotherapy. This type of treatment has been more effective for other types of cancer in the abdomen. Researchers want to see this if approach can improve the outcomes of people with ACC.

Objectives:

- To test the safety and effectiveness of surgery and heated chemotherapy for ACC.

Eligibility:

- Individuals at least 18 years of age who have advanced ACC.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Heart function tests will be given. Imaging studies will be used to locate the surgical sites before the operation.
* Participants will have surgery to remove ACC tumor tissue. After the tumors have been removed, they will have heated chemotherapy with cisplatin. The heat may help weaken any remaining cancer cells and make them easier to destroy. It will also focus the treatment on the tumor sites, rather than the whole body.
* Participants will recover in the hospital for several days after surgery. They will have regular follow-up visits to monitor the outcome of the surgery.

DETAILED DESCRIPTION:
Background:

* Adrenocortical carcinoma (ACC) is a rare tumor with an incidence of 1.5 to 2 per million people per year and has a very poor prognosis with an overall 5-year mortality rate of 75 - 90% and an average survival from the time of diagnosis of 14.5 months.
* The treatment of choice for a localized primary or recurrent tumor is surgical resection. For unresectable metastatic or recurrent disease, mitotane, aminoglutethimide, metapyrone, and ketoconazole are used.
* Cisplatin is one of the most effective chemotherapeutic agents for ACC. In the Surgery Branch we have conducted Phase I and II trials using heated intraperitoneal (IP) chemotherapy with cisplatin for primary peritoneal mesothelioma, low grade appendiceal adenocarcinoma, ovarian malignancies, and high grade adenocarcinoma of the gastrointestinal tract. Synergy has been demonstrated for cisplatin and hyperthermia.
* The purpose of this trial is to determine if an aggressive surgical approach with intraperitoneal administration of heated cisplatin when tumor volume is minimal, can impact and improve on progression free survival.

Objectives:

- To determine IP progression free survival after optimal debulking and heated IP chemotherapy with cisplatin in patients with IP spread of adrenocortical cancer

Eligibility:

- Histologically proven ACC evaluable by computed tomography (CT) imaging with the majority of disease confined to the peritoneal cavity and surgically resectable to a residual size of less than 1 cm or amenable to radiofrequency ablation in patients who are > 18 years of age.

Design:

- This is a classic phase 2 trial to determine efficacy of this therapeutic strategy in ACC. Patients will undergo cytoreductive surgery to achieve a CCR of 0 or 1.

Patients who are successfully debulked will then undergo hyperthermic intraperitoneal chemotherapy (HIPEC) with cisplatin.

Patients will be evaluated by associate investigators in coordination with the Principal Investigator for eligibility. Due to its exploratory nature, up to 30 patients may be enrolled to obtain 24 evaluable patients. (Patients must undergo successful debulking and HIPEC to be considered evaluable.)

ELIGIBILITY:
* INCLUSION CRITERIA
* Histologically proven Adrenocortical carcinoma (ACC) with the majority of disease confined to the peritoneal cavity and resectable or amenable to radiofrequency ablation
* Disease evaluable by computed tomography (CT) or positron emission tomography (PET) imaging
* All disease should be deemed resectable based on imaging studies e.g.:

  * Hepatic metastases (unilateral or bilateral less than or equal to 5 lesions, less than or equal to 15 cm total diameter)
  * Note: Hepatic lesions must be amenable to complete resection
  * Primary peritoneal metastases (small disease load less than or equal to P2 disease) without massive ascites or intestinal obstruction
  * Lung metastases (less than or equal to 3 unilateral/bilateral, 9 cm total diameter)
  * Note: lung lesions must be amenable to complete resection
  * Note: Patients with both pulmonary and hepatic metastases will be enrolled at the discretion of the principal investigator (PI)
  * Note: In situations where resection to Completeness of Cytoreduction Score (CC) 0 or 1 is uncertain, patients may undergo diagnostic laparoscopy prior to enrollment to determine feasibility of resection.
* Greater than or equal to 18 years of age
* Able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy
* Hematology:

  * Absolute neutrophil count greater than 1500/mm^3 without the support of Filgrastim.
  * Platelet count greater than 75,000/mm^3.
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum creatinine less than or equal to 1.5 mg/dl unless the measured creatinine clearance is greater than 60 mL/min/1.73 m2
  * serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within 5 times the upper limit of normal and a total serum bilirubin of less than 3 times the upper limit of normal, both of which define the upper limit of grade 2 treatment related toxicities.
  * Prothrombin time (PT) within 2 seconds of the upper limit of normal (international normalized ratio (INR) less than or equal to 1.8)
* Recovered from any toxicity to grade 2 or less from all prior chemotherapy, immunotherapy or radiotherapy and be at least 30 days past the date of their last treatment with the exception of mitotane which may be continued.
* Able to understand their disease and the exploratory nature of combining surgery and Heated Intraperitoneal Peritoneal Chemotherapy (HIPEC) for this histology.

EXCLUSION CRITERIA

* Concomitant medical problems that would place the patient at unacceptable risk for a major surgical procedure.
* History of congestive heart failure and/or an left ventricular ejection fraction (LVEF) less than 40%

Note: Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., greater than 65yo, diabetes, history of hypertension, elevated low-density lipoproteins (LDL), first degree relative with coronary artery disease) will undergo full cardiac evaluation and will not be eligible if they demonstrate significant irreversible ischemia on stress thallium or an ejection fraction less than 40%.

- Significant Chronic Obstructive Pulmonary Disease (COPD) or other chronic pulmonary restrictive disease with pulmonary function test (PFTs) indicating an forced expiratory volume 1 (FEV1) less than 50% or a Carbon monoxide diffusing capacity (DLCO) less than 40% predicted for age

Note: Patients who have shortness of breath with minimal exertion or who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing and will not be eligible if their FEV1 is less than 50% of expected.

* Grade 2 or greater neuropathy
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
* Brain metastases or a history of brain metastases
* Childs B or C cirrhosis
* Evidence of severe portal hypertension by history, endoscopy, or radiologic studies

Note: Any diagnosis of portal hypertension or clinical stigmata of such including but not limited to gastric or esophageal varices, umbilical vein varices or telangiectasias.

* Weight less than 30 kg
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04-12 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy L Davis, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Datrice NM, Langan RC, Ripley RT, Kemp CD, Steinberg SM, Wood BJ, Libutti SK, Fojo T, Schrump DS, Avital I. Operative management for recurrent and metastatic adrenocortical carcinoma. J Surg Oncol. 2012 Jun 1;105(7):709-13. doi: 10.1002/jso.23015. Epub 2011 Dec 20. PMID 22189845
- [Background] Leboulleux S, Deandreis D, Al Ghuzlan A, Auperin A, Goere D, Dromain C, Elias D, Caillou B, Travagli JP, De Baere T, Lumbroso J, Young J, Schlumberger M, Baudin E. Adrenocortical carcinoma: is the surgical approach a risk factor of peritoneal carcinomatosis? Eur J Endocrinol. 2010 Jun;162(6):1147-53. doi: 10.1530/EJE-09-1096. Epub 2010 Mar 26. PMID 20348273
- [Background] Feldman AL, Libutti SK, Pingpank JF, Bartlett DL, Beresnev TH, Mavroukakis SM, Steinberg SM, Liewehr DJ, Kleiner DE, Alexander HR. Analysis of factors associated with outcome in patients with malignant peritoneal mesothelioma undergoing surgical debulking and intraperitoneal chemotherapy. J Clin Oncol. 2003 Dec 15;21(24):4560-7. doi: 10.1200/JCO.2003.04.150. PMID 14673042
- [Result] Hughes MS, Lo WM, Beresnev T, Merino M, Shutack Y, Ripley RT, Hernandez JM, Davis JL. A Phase II Trial of Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy for Recurrent Adrenocortical Carcinoma. J Surg Res. 2018 Dec;232:383-388. doi: 10.1016/j.jss.2018.06.012. PMID 30463745

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Started | 11
Completed | 10
Not Completed | 1
Not completed — Pt could not be cytoreduced for HIPEC | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.48 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Tumor Stage (AJCC) at Diagnosis [Number; unit: percentage of participants] — American Joint Committee on Cancer (AJCC) - Tumor Stage I-IV with Stage I being the least advanced cancer with the best prognosis, and Stage 4 being the most advanced cancer with the worst prognosis.
  percentage of participants
    Stage I | 20
    Stage II | 50
    Stage III | 10
    Stage IV | 0
    Unknown | 20

OUTCOME MEASURES:

1. Primary Outcome: Intraperitoneal Progression Free Survival (PFS)
Description: Amount of time subject survives without intraperitoneal disease progression after treatment. Disease progression is defined as imageable tumor nodules or increasing ascites persistent on computed tomography (CT) scan as interpreted by the official interpretation of the imaging studies.
Time Frame: Amount of time subject survives without intraperitoneal disease progression after treatment, an average of 17 months
Population: One patient could not be optimally cytoreduced for HIPEC and therefore did not receive intraperitoneal chemotherapy.
Measure: Median (Full Range); unit: Months
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 10
Months | 19 [3 to 66]

2. Secondary Outcome: Number of Patients With Treatment Related Morbidity Following the Heated Intraperitoneal Peritoneal Chemotherapy (HIPEC) Procedure
Description: Patients who died following the HIPEC procedure. The HIPEC is a surgical procedure in which two large bore catheters are inserted in the abdominal wall over the liver and pelvis. The physician closes the abdominal fascia and the catheters are connected to a perfusion circuit. The temperature of the catheters is carefully monitored while the physician ensures the perfusion is distributed properly by manually moving the abdomen.
Time Frame: Patients were assessed every 3 months up to an average of 17 months.
Population: One patient could not be optimally cytoreduced for HIPEC and therefore did not receive intraperitoneal chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Percentage of Participants Who Survived 5-years Post Treatment
Description: Percentage of participants who are alive after treatment.
Time Frame: 5 years
Population: Nine patients underwent cytoreduction and HIPEC, including one patient who recurred and was re-treated (n = 10 treatments). One patient could not be optimally cytoreduced for HIPEC and therefore did not receive intraperitoneal chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 9
percentage of participants | 66.7 [28.2 to 87.8]

4. Secondary Outcome: The Functional Assessment of Cancer Therapy-Colorectal Quality of Life (FACT-G) (QOL) Score Prior to Surgery, 6 Weeks After Surgery, and 3 Months After Surgery
Description: QOL characteristics were collected using The Functional Assessment of Cancer Therapy-Colorectal Quality of Life (QOL) questionnaire version 4, a validated survey that interrogates physical, emotional, functional, and social well being in cancer related issues on a 5-point scale. Scores range from 0 to 108 points. Higher scores are consistent with a better outcome.
Time Frame: Prior to surgery, 6 weeks post surgery, and 3 months post surgery
Population: One patient could not be optimally cytoreduced for hyperthermic intraperitoneal chemotherapy (HIPEC) and therefore did not receive intraperitoneal chemotherapy.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 11
scores on a scale
  Prior to surgery | 82.6 [NA to NA] — The full range data is unavailable because the primary source documents are not available. All of the personnel involved in the running of the study, data acquisition, and the person who put together the manuscript have all left the NIH.
  6 weeks after surgery | 76.4 [NA to NA] — The full range data is unavailable because the primary source documents are not available. All of the personnel involved in the running of the study, data acquisition, and the person who put together the manuscript have all left the NIH.
  3 months after surgery | 80.2 [NA to NA] — The full range data is unavailable because the primary source documents are not available. All of the personnel involved in the running of the study, data acquisition, and the person who put together the manuscript have all left the NIH.

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytoreductive Surgery Followed by HIPEC
Number analyzed (Participants) | 11
Participants | 8

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 28 days.
Arm/Group | Cytoreductive Surgery Followed by HIPEC
All-Cause Mortality (participants affected / at risk) | 3/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytoreductive Surgery Followed by HIPEC (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytoreductive Surgery Followed by HIPEC (N=11)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Platelet count decreased (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT01833832/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT01833832/ICF_001.pdf